CLINICAL TRIAL: NCT01748890
Title: A Pilot Trial of Sonoelastography for Planning Tumor-targeted Prostate Biopsy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Anthony Samir, Assistant Radiologist, Ultrasound Imaging Services Assistant Radiologist, Abdominal Imaging & Intervention, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-395
Record Dates: First submitted 2012-10-31; First posted 2012-12-13 (Estimated); Results first posted 2014-05-20 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sonoelastography (Experimental): Sonoelastography is an imaging technology predicated on reproducible differences in the backscattered ultrasound signal produced by compression of tissues of varying stiffness.
  Interventions: Device: Sonoelastography

INTERVENTIONS:
Device: Sonoelastography — Sonoelastography is an imaging technology predicated on reproducible differences in the backscattered ultrasound signal produced by compression of tissues of varying stiffness.
  Other Names: Hitachi; HI VISION Preirus

SUMMARY:
Prostate cancer is the most common cancer and the second-leading cause of cancer death amongst men in the United States. Sonoelastography is an imaging technology predicated on reproducible differences in the backscattered ultrasound signal produced by compression of tissues of varying stiffness. It permits measurement of the elastic properties of tissue. These measurements can be transposed onto conventional anatomic ultrasound images, producing a colorized overlay that allows direct visualization of the anatomic distribution of tissue stiffness. In this study, we aim to determine whether prostate biopsies planned with sonoelastographic guidance would be more likely than random prostate biopsies to intersect with foci of carcinoma in the prostate gland, and to determine whether prostate biopsies planned with sonoelastographic guidance would be more likely than random prostate biopsies to yield histopathology representative of the final Gleason Score obtained at pathologic assessment of the resected prostate.

DETAILED DESCRIPTION:
Background and Significance Prostate cancer is the most common cancer and the second-leading cause of cancer death amongst men in the United States. Initially, tumors biopsy guided by detected by conventional B-mode transrectal ultrasound (TRUS). Unfortunately, prostate cancer had a highly variable ultrasound echo pattern and may be indistinguishable from normal prostate, and the sonographic appearance of BPH overlaps with that of prostatic carcinoma, which limited the accuracy of conventional ultrasound, producing sensitivity and specificity for prostate carcinoma of only 40-50%. There is therefore an urgent need for better localization and more accurate biopsy of prostate cancer.

Sonoelastography is an imaging technology predicated on reproducible differences in the backscattered ultrasound signal produced by compression of tissues of varying stiffness. It permits measurement of the elastic properties of tissue. These measurements can be transposed onto conventional anatomic ultrasound images, producing a colorized overlay that allows direct visualization of the anatomic distribution of tissue stiffness.

Previously, several studies have reported that the feasibility of sonoelastography to distinguish between benign and malignant nodules and thereby guide biopsy. These assessments were based on the change in anatomic appearance of nodules after compression with a transrectal ultrasound probe. However, these reports did not specify the criteria used to determine that lesions seen by elastography were the same lesions seen by histopathology, did not assess whether biopsies planned with the assistance of sonoelastography would have intersected with the foci of prostate cancer, and did not address the histopathologic characteristics of areas of the prostate that were falsely positive at sonoelastography.

If sonoelastography were to more accurately delineate foci of tumor in the prostate than B mode ultrasound, and it could be used to guide biopsy, then there would be fewer missed cancers at biopsy. In addition, sonoelastography-guided biopsies may be more representative of the ultimate Gleason Score of the tumor.

Specific Aims:

Aim 1: To determine whether prostate biopsies planned with sonoelastographic guidance would be more likely than random prostate biopsies to intersect with foci of carcinoma in the prostate gland.

Aim 2: To determine whether prostate biopsies planned with sonoelastographic guidance would be more likely than random prostate biopsies to yield histopathology representative of the final Gleason Score obtained at pathologic assessment of the resected prostate.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years of age or older.
2. Serum PSA between 4 and 10 ng/mL.
3. A diagnosis of prostate cancer based on extended (twelve core) random prostate biopsy within three months prior to study entry.
4. Clinically localized prostate carcinoma i.e. TNM stage T2c or less.
5. The patient has elected to undergo radical prostatectomy to treat the prostate carcinoma.
6. The patient consents to undergo a diagnostic transrectal ultrasound of the prostate with elastography.

Exclusion Criteria:

1. Any contraindication to transrectal ultrasonography, including prior anorectal surgery, inflammatory bowel disease, rectal fistula, or fissure-in-ano.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony E. Samir, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sonoelastography
Started | 4
Completed | 0 (Insufficient recruitment for analysis)
Not Completed | 4
Not completed — Insufficient recruitment for analysis | 4

BASELINE CHARACTERISTICS:
Arm/Group | Sonoelastography
Number analyzed (Participants) | 0
Age, Continuous [unit: years]
Age, Categorical
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: The Number of Core Biopsies in These Targeted Regions
Description: From elastography-prostatectomy pathology correlation, the following data will be obtained, 1) The number of planned core biopsies that would intersect foci of prostate carcinoma, 2) The Gleason Score that would be obtained, assuming that elastographically targeted biopsies sample the targeted region.
Time Frame: Participants will be followed until prostatectomy pathology is available (average 1 week)
Population: insufficient recruitment for analysis
Arm/Group | Sonoelastography
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The adverse event data were monitored and collected every 6 months.
Description: No adverse event was found to date.
Arm/Group | Sonoelastography
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes